CLINICAL TRIAL: NCT00251706
Title: Prophylactic Amiodarone for the Prevention of Arrhythmias That Begin Early After Revascularization, Valve Replacement, or Repair - PAPABEAR
Brief Title: Amiodarone to Prevent Post-Operative Arrhythmias
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Heart and Stroke Foundation of Canada (Other); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PAPABEAR; CIHR MCT-14764
Record Dates: First submitted 2005-11-08; First posted 2005-11-10 (Estimated); Last update posted 2006-05-05 (Estimated); Status verified 2005-11

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; atrial flutter; amiodarone; post-operative; coronary artery bypass surgery; valve replacement or repair
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter | interventions — Amiodarone

INTERVENTIONS:
Drug: amiodarone

SUMMARY:
Rapid heart rhythms originating from the upper heart chambers (atrial tachyarrhythmias) are very common after open-heart surgery. The hypothesis of the PAPABEAR study is that a brief (13 day) peri-operative course of oral amiodarone therapy would be effective and safe for the prevention of these post-operative atrial tachyarrhythmias.

DETAILED DESCRIPTION:
Six hundred and one patients who were about to undergo non-emergent open-heart surgery were randomized to receive oral amiodarone (10 mg/kg/day) or its matching placebo from six days before surgery through 6 days after surgery. The major outcome tracked was the incidence of more than 5 minutes of an atrial tachyarrhythmia that prompted therapy by the sixth post-operative day. Safety was assessed by the incidence of dosage reduction of blinded therapy, non-fatal post-operative complications, and in-hospital mortality. The randomization scheme was stratified to permit separate analysis of patients less than versus more than or equal to 65 years of age, patients having coronary artery bypass surgery alone versus those having valve surgery with or without concomitant bypass surgery, and patients also receiving versus not also receiving concomitant therapy with a beta-blocker medication.

ELIGIBILITY:
Inclusion Criteria:

* non-emergent coronary artery bypass surgery or valve replacement or repair
* informed consent

Exclusion Criteria:

* any heart rhythm other than sinus
* myocardial infarction within two weeks
* Class IV congestive Heart Failure
* requirement for antiarrhythmic drug therapy
* history of sustained atrial tachyarrhythmias
* treatment with amiodarone within 3 months
* sinus bradycardia (less than 50 bpm) while awake
* advanced conduction system disease
* prolonged QT interval
* clinical hypo- or hyperthyroidism
* women of child bearing potential

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600
Dates: Start 1999-02; Study Completion 2004-09

PRIMARY OUTCOMES:
more than 5 minutes of post-operative atrial tachyarrhythmia
ventricular response rate of atrial tachyarrhythmias
burden of post-operate atrial tachyarrhythmias
length of hospital stay

SECONDARY OUTCOMES:
withdrawal of full-dose blinded therapy
non-fatal post-operative complications
hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: L. Brent Mitchell, MD, Principal Investigator — University of Calgary
Locations (1):
- Libin Cardiovascular Institute / University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Result] Mitchell LB, Exner DV, Wyse DG, Connolly CJ, Prystai GD, Bayes AJ, Kidd WT, Kieser T, Burgess JJ, Ferland A, MacAdams CL, Maitland A. Prophylactic Oral Amiodarone for the Prevention of Arrhythmias that Begin Early After Revascularization, Valve Replacement, or Repair: PAPABEAR: a randomized controlled trial. JAMA. 2005 Dec 28;294(24):3093-100. doi: 10.1001/jama.294.24.3093. PMID 16380589